CLINICAL TRIAL: NCT05160766
Title: A Multinational, Phase 2, Randomised, Adaptive Protocol to Evaluate Immunogenicity and Reactogenicity of Different COVID-19 Vaccines Administration in Older Adults (≥75) Already Vaccinated Against SARS-COV-2 (EU-COVAT-1_AGED)
Brief Title: Assessing Immune Response of Different COVID-19 Vaccines in Older Adults
Acronym: EU-COVAT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oliver Cornely, MD (Other)
Collaborators: VACCELERATE (Unknown); European Commission (Other)
Responsible Party: Sponsor-Investigator, Oliver Cornely, MD, Principal Coordinating Investigator, University of Cologne
Organization: University of Cologne (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EU-COVAT-1_AGED; 2021-004526-29 (EudraCT Number); uni-koeln-4602 (Other: University of Cologne)
Record Dates: First submitted 2021-11-11; First posted 2021-12-16 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Prevention of COVID-19
Keywords: SARS-CoV-2; COVID-19; Vaccination; Immunogenicity; BNT162b2; mRNA-1273; Booster; Elderly; head-to-head comparison
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: This is a randomised controlled, adaptive, multicentre Phase II protocol evaluating different booster strategies in individuals aged 75 years and older already vaccinated against SARS-CoV-2. This trial foresees testing of different vaccines as a third (first booster, Part A) or fourth vaccine dose (second booster, Part B) for comparative assessment of their immunogenicity and safety against SARS-CoV-2 and SARS-CoV-2 variants in the elderly.
Masking Description: No blinding is foreseen in this trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- BNT162b2 (Part A) (Active Comparator): vaccination with BNT162b2 as 3rd vaccination
  Interventions: Biological: Comirnaty (BTN162b2)
- mRNA-1273 (Part A) (Active Comparator): vaccination with mRNA-1273 as 3rd vaccination
  Interventions: Biological: Spikevax (mRNA-1273)
- BNT162b2 (Part B) (Active Comparator): vaccination with BNT162b2 as 4th vaccination
  Interventions: Biological: Comirnaty (BTN162b2)
- mRNA-1273 (Part B) (Active Comparator): vaccination with mRNA-1273 as 4th vaccination
  Interventions: Biological: Spikevax (mRNA-1273)

INTERVENTIONS:
Biological: Comirnaty (BTN162b2) — Single booster shot (3rd dose in Part A and 4th dose in Part B)
  Arms: BNT162b2 (Part A); BNT162b2 (Part B)
Biological: Spikevax (mRNA-1273) — Single booster shot (3rd dose in Part A and 4th dose in Part B)
  Arms: mRNA-1273 (Part A); mRNA-1273 (Part B)

SUMMARY:
This is a randomised controlled, adaptive, multicentre Phase II protocol evaluating different booster strategies in individuals aged 75 years and older already vaccinated against SARS-CoV-2.

Part A of this trial foresees testing of different vaccines as a 3rd vaccination dose (first booster) for comparative assessment of their immunogenicity and safety against SARS-CoV-2 wild-type and variants in the elderly, a usually neglected population.

Part B of this trial foresees testing of different vaccines as a 4th vaccination dose (second booster) for comparative assessment of their immunogenicity and safety against SARSCoV-2 wild-type and variants in the identical population.

DETAILED DESCRIPTION:
Part A of the present trial in which individuals received a 3rd vaccination (first booster) of either BNT162b2 or mRNA-1273 was closed to further recruitment as of January 13, 2022. This was due to a change in vaccination policies, recommending a 3rd vaccination with either BNT162b2 or mRNA-1273. Therefore, Part A was supplanted by Part B that investigated a 4th COVID-19 vaccination and started on 21 Jan 2022.

The initial study protocol started the trial with Part A in which participants were randomized to a 3rd vaccination (first booster) with either BNT162b2 or mRNA-1273:

Subjects who - prior to study entry - received a vaccination series of either BNT162b2 & BNT162b2 or mRNA-1273 & mRNA-1273 or ChAdOx-1-S & ChAdOx-1-S.

For the reasons mentioned above, the study protocol was amended to continue the trial with Part B in which participants were randomized to a 4th vaccination (second booster) with either BNT162b2 or mRNA-1273:

Subjects who - prior to study entry - received a vaccination series of either BNT162b2 & BNT162b2 & BNT162b2 or BNT162b2 & BNT162b2 & mRNA-1273 or mRNA-1273 & mRNA-1273 & mRNA-1273 or mRNA-1273 & mRNA-1273 & BNT162b2 or ChAdOx-1-S & ChAdOx-1-S & BNT162b2 or ChAdOx-1-S & ChAdOx-1-S & mRNA-1273.

ELIGIBILITY:
Inclusion Criteria (Part A):

* Subject is ≥75 years old.
* Prior to study entry the subject was vaccinated with BNT162b2, mRNA-1273 or ChAdOx-1-S (same vaccine product for 1st + 2nd dose)

BNT162b2 + BNT162b2

mRNA-1273 + mRNA-1273

ChAdOx-1-S + ChAdOx-1-S

* 9 ± 3 months since the second vaccine dose at time of enrolment for the planned 3rd vaccine dose in the trial. Vaccination status should be documented in the source data and captured in the eCRF.
* No contra-indication against any of the vaccine products in the trial.
* Written informed consent from subject has been obtained.

Exclusion Criteria (Part A):

* Primary vaccination performed with different vaccine products as sole (e.g., COVID-19 Vaccine Janssen) or, 1st and 2nd vaccination doses (heterologous vaccination scheme).
* Subjects with any significant or uncontrolled disease posing a risk due to vaccination as judged by the investigator.
* Current immunosuppressive therapy, for example continuous glucocorticosteroid treatment equivalent to >10 mg/day prednisolone.
* Participation in other interventional trials.
* Subjects unable to report solicited adverse events.
* Subject with any contraindications to the vaccines in the trial at randomisation. A list of contraindications as listed in the Summary of medicinal Product Characteristics (SmPC, the Fachinformation in Germany), if appropriate.
* Use of drugs with significant interaction with the investigational product according to the SmPC or similar documents.
* Diseases or findings that may have a significant effect on the target variables and which may therefore mask or inhibit the therapeutic effect under investigation.
* Any current SARS-CoV-2 infection or proven in the preceding 3 months.
* Persons with any kind of dependency on the principal investigator or employed by the sponsor or principal investigator.
* Legally incapacitated persons.
* Persons held in an institution by legal or official order.

Inclusion Criteria (Part B):

* Subject is ≥75 years old.
* Prior to study entry the subject was vaccinated with one of the following vaccination regimens (1st + 2nd + 3rd dose):

BNT162b2 + BNT162b2 + BNT162b2

BNT162b2 + BNT162b2 + mRNA-1273

mRNA-1273 + mRNA-1273 + mRNA-1273

mRNA-1273 + mRNA-1273 + BNT162b2

ChAdOx-1-S + ChAdOx-1-S + BNT162b2

ChAdOx-1-S + ChAdOx-1-S + mRNA-1273

The last dose of the above listed vaccinations must have been administered at least 1 month prior to study entry. Vaccination status should be documented in the source data and will be captured in the eCRF.

- Written informed consent from subject has been obtained.

Exclusion Criteria (Part B):

* Prior to study entry the subject got vaccinated with a regimen not included in the list given above.
* Last anti-SARS-CoV-2 vaccine dose administered less than one month prior to study entry.
* Vaccination against a disease other than COVID-19 within 2 weeks prior to study entry. Only exception: Influenza vaccination which is allowed at any time.
* Subjects with any significant or uncontrolled disease posing a risk due to vaccination as judged by the investigator.
* Current immunosuppressive therapy, for example continuous glucocorticosteroid treatment equivalent to >10 mg/day prednisolone.
* Subject simultaneously participates in another clinical trials or has participated in the past 30 days.
* Subjects unable to report solicited adverse events.
* Subject with any contraindications to the vaccines in the trial. A list of contraindications as listed in the Summary of medicinal Product Characteristics (SmPC, the Fachinformation in Germany), if appropriate.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 323 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A Cornely, MD, Principal Investigator — University of Cologne
Locations (9):
- Germany (3):
  - University Hospital Cologne, Cologne
  - University Hospital Frankfurt, Frankfurt
  - Hannover Medical School Hospital, Hanover
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Helse Bergen HF, Haukeland University Hospital, Bergen, Norway
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Reina Sofia University Hospital, Córdoba
  - La Paz University Hospital, Madrid
  - Biodonostia Health Research Institute, San Sebastián

IPD SHARING:
Plan to Share IPD: Yes
Making de-identified/anonymized data accessible is currently under way. We expect to grant access through a central independent data repository no later than January 2025. Any pertinent information will be updated in due course.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Making de-identified/anonymized data accessible is currently under way. We expect to grant access through a central independent data repository no later than January 2025. Any pertinent information will be updated in due course.
Access Criteria: To be announced.

REFERENCES:
- [Derived] Neuhann JM, Stemler J, Carcas A, Frias-Iniesta J, Bethe U, Heringer S, Tischmann L, Zarrouk M, Cuppers A, Konig F, Posch M, Cornely OA. A multinational, phase 2, randomised, adaptive protocol to evaluate immunogenicity and reactogenicity of different COVID-19 vaccines in adults >/=75 already vaccinated against SARS-CoV-2 (EU-COVAT-1-AGED): a trial conducted within the VACCELERATE network. Trials. 2022 Oct 8;23(1):865. doi: 10.1186/s13063-022-06791-y. PMID 36209129

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to poor recruitment, Part A of the trial (3rd COVID-19 vaccination) was closed to further enrolment on 13 Jan 2022. Part B (4th COVID-19 vaccination) started on 21 Jan 2022.
  In Part A, one randomised subject did not receive the allocated intervention (mRNA-1273) due to an acute onset of SARS-CoV-2 infection.
  Both Part A and B belong to one trial and fall under one NCT number.
Groups:
- BNT162b2 (Part A); mRNA-1273 (Part A): Part A:
  Participants were pre-vaccinated with 2 vaccinations when entering the trial, as follows:
  BNT162b2 + BNT162b2 mRNA-1273 + mRNA-1273 ChAdOx-1-S + ChAdOx-1-S
  A 3rd dose was administered in the study, either Comirnaty (BTN162b2) or Spikevax (mRNA-1273).
- BTN162b2 (Part B); mRNA-1273 (Part B): Part B:
  Participants were pre-vaccinated with 3 vaccinations when entering the trial, as follows:
  BNT162b2 + BNT162b2 + BNT162b2 BNT162b2 + BNT162b2 + mRNA-1273 mRNA-1273 + mRNA-1273 + mRNA-1273 mRNA-1273 + mRNA-1273 + BNT162b2 ChAdOx-1-S + ChAdOx-1-S + BNT162b2 ChAdOx-1-S + ChAdOx-1-S + mRNA-1273
  A 4th dose was administered in the study, either Comirnaty (BTN162b2) or Spikevax (mRNA-1273).
Period: Overall Study
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BTN162b2 (Part B) | mRNA-1273 (Part B)
Started | 25 | 27 | 135 | 135
Completed | 21 | 20 | 126 | 123
Not Completed | 4 | 7 | 9 | 12
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — COVID-19 infection | 0 | 1 | 0 | 0
Not completed — travel time | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 4 | 2
Not completed — Death | 0 | 0 | 2 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1 | 2
Not completed — No show | 0 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- BNT162b2 (Part B); mRNA-1273 (Part B): Part B:
  Participants were pre-vaccinated with 3 vaccinations when entering the trial, as follows:
  BNT162b2 + BNT162b2 + BNT162b2 BNT162b2 + BNT162b2 + mRNA-1273 mRNA-1273 + mRNA-1273 + mRNA-1273 mRNA-1273 + mRNA-1273 + BNT162b2 ChAdOx-1-S + ChAdOx-1-S + BNT162b2 ChAdOx-1-S + ChAdOx-1-S + mRNA-1273 A 4th dose was administered in the study, either Comirnaty (BTN162b2) or Spikevax (mRNA-1273).
- Total: Total of all reporting groups
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B) | Total
Number analyzed (Participants) | 25 | 27 | 135 | 135 | 322
Age, Continuous [Median (Full Range); unit: years] | 77 [75 to 87] | 78 [75 to 85] | 79 [75 to 99] | 79 [75 to 99] | 79 [75 to 99]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 67 | 68 | 155
  Male | 16 | 16 | 68 | 67 | 167
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Median (Full Range); unit: cm] | 171 [155 to 190] | 174 [149 to 198] | 169 [143 to 189] | 169 [145 to 198] | 169 [143 to 198]
Weight [Median (Full Range); unit: kg] | 75 [53 to 97] | 73 [51 to 100] | 72 [41 to 119] | 75 [41.7 to 110] | 74 [41 to 119]
BMI [Median (Full Range); unit: kg/m2] | 25.6 [20.3 to 32.8] | 24.1 [16.8 to 32.6] | 25.4 [16.6 to 40.2] | 25.4 [18 to 41.8] | 25.4 [16.6 to 41.8]
Duration between 1st and 2nd vaccination in days [Median (Full Range); unit: days] | 42 [21 to 84] | 42 [21 to 111] | 22 [20 to 86] | 22 [16 to 114] | 22 [16 to 114]
Duration between 2nd and 3rd vaccination in days [Median (Full Range); unit: days] | 192 [185 to 255] | 190 [184 to 273] | 207 [124 to 303] | 205 [126 to 313] | 206.5 [124 to 313]

OUTCOME MEASURES:

1. Primary Outcome: Antibody Titre Increase 14 Days After Study Vaccination Dose.
Description: Rate of 2-fold antibody titre increase 14 days after 3rd (Part A) or 4th vaccination dose (Part B) measured by qualitative enzyme-linked immunosorbent assay (Anti-RBD-ELISA) against wildtype virus.
Time Frame: From Day 0 until Day 14
Population: All primary analyses were performed on the mITT population set. The primary endpoint was the rate π of 2-fold IgG antibody titre increase following a 3rd (Part A) or 4th dose vaccination (Part B) measured by quantitative enzyme-linked electrochemiluminescent immunoassay (Anti-RBD-ELISA) against wild-type virus at 14 days after study vaccination (versus immediately before vaccination).
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Groups:
- BNT162b2 (Part A): vaccination with BNT162b2 as 3rd vaccination
  Comirnaty (BTN162b2): Single booster shot (3rd dose)
- mRNA-1273 (Part A): vaccination with mRNA-1273 as 3rd vaccination
  Spikevax (mRNA-1273): Single booster shot (3rd dose)
- BNT162b2 (Part B): vaccination with BNT162b2 as 4th vaccination
  Comirnaty (BTN162b2): Single booster shot (4th dose)
- mRNA-1273 (Part B): vaccination with mRNA-1273 as 4th vaccination
  Spikevax (mRNA-1273): Single booster shot (4th dose)
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B)
Number analyzed (Participants) | 25 | 25 | 130 | 133
percentage of participants | 100 [83.9 to 100] | 100 [83.9 to 100] | 78.46 [69.2 to 86] | 87.22 [79.3 to 93]

2. Secondary Outcome: Change in Neutralizing Antibody Titre Against Wild-type 14 Days After Study Vaccination Dose
Description: Change in neutralizing antibody titre (Virus Neutralisation Assay) against wild-type 14 days after a 3rd (Part A) or 4th vaccination dose (Part B), to be determined in a subgroup only.
  Microneutralization assay results were proposed to be reported as "change in neutralizing antibody titre (Virus Neutralisation Assay)" in the trial protocol. However, as the pandemic progressed, the need arose to assess neutralization against different variants. In our stud(ies), we evaluated not only the Wuhan strain but also 25 distinct variants of concern (VoCs) and/or variants of interest (VoIs). For VoCs and VoIs, expressing results as "change in neutralization capacity expressed as a percentage (%)" is more effective as it illustrates the impact of mutations on neutralization, thereby allowing cross-variant comparisons. This adjustment did not alter the suggested endpoint, as both reporting methods reflect the ability of patients' antibodies neutralizing capacities.
Time Frame: From Day 0 until Day 14
Population: Number of subjects for whom the difference of neutralizing activity (Day 14 minus Day 0) could be calculated.
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Groups:
- BTN162b2 (Part A): vaccination with BNT162b2 as 3rd vaccination
  Comirnaty (BTN162b2): Single booster shot (3rd dose)
- BTN162b2 (Part B): vaccination with BNT162b2 as 4th vaccination
  Comirnaty (BTN162b2): Single booster shot (4th dose)
Arm/Group | BTN162b2 (Part A) | mRNA-1273 (Part A) | BTN162b2 (Part B) | mRNA-1273 (Part B)
Number analyzed (Participants) | 21 | 20 | 122 | 120
percentage of inhibition | 58.49 (16.25) | 65.98 (18.32) | 37.33 (22.93) | 41.45 (24.09)
Statistical Analysis 1: Comparison: BTN162b2 (Part A) vs mRNA-1273 (Part A); The statistical analysis reflects Part A of the study; Test type: Other; p = 0.03143, ANCOVA; Difference of means in percent = 12.557, 95% CI 2-sided [1.168 to 23.946], Standard Error of Mean 5.661
Statistical Analysis 2: Comparison: BTN162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.0101, ANCOVA; Difference of means in percent = 4.331, 95% CI 2-sided [1.04 to 7.621], Standard Error of Mean 1.671

3. Secondary Outcome: Change in Neutralizing Antibody Titre Against Variants of Concern 14 Days After Study Vaccination Dose
Description: Change in neutralizing antibody titre (Virus Neutralisation Assay) against variants of concern 14 days after a 3rd (Part A) or 4th vaccination dose (Part B), to be determined in a subgroup only.
  Microneutralization assay results were proposed to be reported as "change in neutralizing antibody titre (Virus Neutralisation Assay)" in the trial protocol. However, as the pandemic progressed, the need arose to assess neutralization against different variants. In our stud(ies), we evaluated not only the Wuhan strain but also 25 distinct variants of concern (VoCs) and/or variants of interest (VoIs). For VoCs and VoIs, expressing results as "change in neutralization capacity expressed as a percentage (%)" is more effective as it illustrates the impact of mutations on neutralization, thereby allowing cross-variant comparisons. This adjustment did not alter the suggested endpoint, as both reporting methods reflect the ability of patients' antibodies neutralizing capacities.
Time Frame: From Day 0 until Day 14
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B)
Number analyzed (Participants) | 21 | 20 | 122 | 120
percentage of inhibition | 49.86 (17.62) | 57.39 (19.77) | 38.17 (21.74) | 44.04 (23.94)
Statistical Analysis 1: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.04405, ANCOVA; Difference of means in percent = 12.168, 95% CI 2-sided [0.338 to 23.998], Standard Error of Mean 5.88; The above provided values refer to the variant "B.1.1.7 (alpha)"
Statistical Analysis 2: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.01744, ANCOVA; Difference of means in percent = 14.212, 95% CI 2-sided [2.61 to 25.814], Standard Error of Mean 5.767; The above provided values refer to the variant "B.1.351 (beta)"
Statistical Analysis 3: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.02039, ANCOVA; Difference of means in percent = 14.239, 95% CI 2-sided [2.305 to 26.173], Standard Error of Mean 5.932; The above provided values refer to the variant "P.1 (gamma)"
Statistical Analysis 4: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.04989, ANCOVA; Difference of means in percent = 9.331, 95% CI 2-sided [0.005 to 18.656], Standard Error of Mean 4.636; The above provided values refer to the variant "BA.1 (omicron)"
Statistical Analysis 5: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.02259, ANCOVA; Difference of means in percent = 10.312, 95% CI 2-sided [1.514 to 19.111], Standard Error of Mean 4.373; The above provided values refer to the variant "BA.4 (omicron)"
Statistical Analysis 6: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.01583, ANCOVA; Difference of means in percent = 11.601, 95% CI 2-sided [2.279 to 20.924], Standard Error of Mean 4.634; The above provided values refer to the variant "BA.4.6 (omicron)"
Statistical Analysis 7: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.00856, ANCOVA; Difference of means in percent = 11.863, 95% CI 2-sided [3.166 to 20.56], Standard Error of Mean 4.323; The above provided values refer to the variant "BA.5 (omicron)"
Statistical Analysis 8: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.00258, ANCOVA; Difference of means in percent = 6.83, 95% CI 2-sided [2.41 to 11.249], Standard Error of Mean 2.244; The above provided values refer to the variant "B.1.1.7 (alpha)"
Statistical Analysis 9: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.00748, ANCOVA; Difference of means in percent = 6.048, 95% CI 2-sided [1.63 to 10.466], Standard Error of Mean 2.244; The above provided values refer to the variant "B.1.351 (beta)"
Statistical Analysis 10: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.00922, ANCOVA; Difference of means in percent = 7.302, 95% CI 2-sided [1.821 to 12.782], Standard Error of Mean 2.782; The above provided values refer to the variant "P.1 (gamma)"
Statistical Analysis 11: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.07136, ANCOVA; Difference of means in percent = 4.791, 95% CI 2-sided [-0.419 to 10.001], Standard Error of Mean 2.646; The above provided values refer to the variant "BA.1 (omicron)"
Statistical Analysis 12: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.07218, ANCOVA; Difference of means in percent = 3.965, 95% CI 2-sided [-0.36 to 8.29], Standard Error of Mean 2.196; The above provided values refer to the variant "BA.4 (omicron)"
Statistical Analysis 13: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.02949, ANCOVA; Difference of means in percent = 4.82, 95% CI 2-sided [0.484 to 9.155], Standard Error of Mean 2.202; The above provided values refer to the variant "BA.4.6 (omicron)"
Statistical Analysis 14: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.08403, ANCOVA; Difference of means in percent = 3.926, 95% CI 2-sided [-0.531 to 8.382], Standard Error of Mean 2.263; The above provided values refer to the variant "BA.5 (omicron)"

4. Secondary Outcome: Antibody Titre Level at 12 Months After a Study Vaccination Dose
Description: Antibody titre level at 12 months after a 3rd (Part A) or 4th vaccination dose (Part B) measured by a quantitative enzyme-linked immunosorbent assay (anti-RBD-ELISA assay).
Time Frame: From Day 0 until Month 12
Population: Subjects in whom a blood sampling was performed at Month 12.
Measure: Geometric Mean (Standard Deviation); unit: IU/ml
Arm/Group | BTN162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B)
Number analyzed (Participants) | 21 | 21 | 125 | 121
IU/ml | 9319.7 (25896.27) | 14163.81 (46209.35) | 9961.92 (26292.23) | 12024.3 (29129.18)

5. Secondary Outcome: Neutralizing Antibody Titre Against Wild-type at 12 Months After Study Vaccination Dose
Description: Neutralizing antibody titre (Virus Neutralisation Assay) against wild-type SARS-CoV-2 at 12 months after a 3rd (Part A) or 4th vaccination dose (Part B), to be determined in a subgroup only.
  Microneutralization assay results were proposed to be reported as "change in neutralizing antibody titre (Virus Neutralisation Assay)" in the trial protocol. However, as the pandemic progressed, the need arose to assess neutralization against different variants. In our stud(ies), we evaluated not only the Wuhan strain but also 25 distinct variants of concern (VoCs) and/or variants of interest (VoIs). For VoCs and VoIs, expressing results as "change in neutralization capacity expressed as a percentage (%)" is more effective as it illustrates the impact of mutations on neutralization, thereby allowing cross-variant comparisons. This adjustment did not alter the suggested endpoint, as both reporting methods reflect the ability of patients' antibodies neutralizing capacities.
Time Frame: From Day 0 until Month 12
Population: Titres of neutralizing antibodies were reported as change in neutralization capacity.
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B)
Number analyzed (Participants) | 21 | 20 | 120 | 120
percentage of inhibition | 54.5 (33.64) | 62.65 (33.26) | 12.93 (39.29) | 18.15 (33.24)

6. Secondary Outcome: Neutralizing Antibody Titre Against Variants of Concern at 12 Months After Study Vaccination Dose
Description: Neutralizing antibody titre (Virus Neutralisation Assay) against variants of concern at 12 months after a 3rd (Part A) or 4th vaccination dose (Part B), to be determined in a subgroup only.
  Microneutralization assay results were proposed to be reported as "change in neutralizing antibody titre (Virus Neutralisation Assay)" in the trial protocol. However, as the pandemic progressed, the need arose to assess neutralization against different variants. In our stud(ies), we evaluated not only the Wuhan strain but also 25 distinct variants of concern (VoCs) and/or variants of interest (VoIs). For VoCs and VoIs, expressing results as "change in neutralization capacity expressed as a percentage (%)" is more effective as it illustrates the impact of mutations on neutralization, thereby allowing cross-variant comparisons. This adjustment did not alter the suggested endpoint, as both reporting methods reflect the ability of patients' antibodies neutralizing capacities.
Time Frame: From Day 0 until Month 12
Population: Titres of neutralizing antibodies were reported as change in neutralization capacity. Provided values refer to the variant "B.1.1.7 (alpha)". Besides for B.1.1.7 (alpha), all tests described above were also conducted for the following variants of concern: B.1.351 (beta), P.1 (gamma), BA.1 (omicron), BA.4 (omicron), BA.4.6 (omicron), and BA.5 (omicron).
  For values of these variants of concern, please see the open-access publication.
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B)
Number analyzed (Participants) | 21 | 20 | 119 | 120
percentage of inhibition | 40.59 (35.37) | 49 (36.37) | 15.76 (38.4) | 20.24 (37.24)
Statistical Analysis 1: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.42797, ANCOVA; Difference of means in percent = 8.835, 95% CI 2-sided [-13.475 to 31.145], Standard Error of Mean 11.03; The above provided values refer to the variant "B.1.1.7 (alpha)"
Statistical Analysis 2: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.73961, ANCOVA; Difference of means in percent = 3.54, 95% CI 2-sided [-17.85 to 24.929], Standard Error of Mean 10.575; The above provided values refer to the variant "B.1.351 (beta)"
Statistical Analysis 3: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.45370, ANCOVA; Difference of means in percent = 8.086, 95% CI 2-sided [-13.524 to 29.695], Standard Error of Mean 10.683; The above provided values refer to the variant "P.1 (gamma)"
Statistical Analysis 4: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.87323, ANCOVA; Difference of means in percent = 1.636, 95% CI 2-sided [-18.969 to 22.241], Standard Error of Mean 10.187; The above provided values refer to the variant "BA.1 (omicron)"
Statistical Analysis 5: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis relfects Part A of the study; Test type: Other; p = 0.93489, ANCOVA; Difference of means in percent = 0.81, 95% CI 2-sided [-19.109 to 20.728], Standard Error of Mean 9.848; The above provided values refer to the variant "BA.4 (omicron)"
Statistical Analysis 6: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.74784, ANCOVA; Difference of means in percent = 3.511, 95% CI 2-sided [-18.425 to 25.448], Standard Error of Mean 10.845; The above provided values refer to the variant "BA.4.6 (omicron)"
Statistical Analysis 7: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.84202, ANCOVA; Difference of means in percent = 2.088, 95% CI 2-sided [-18.966 to 23.143], Standard Error of Mean 10.409; The above provided values refer to the variant "BA.5 (omicron)"
Statistical Analysis 8: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.15477, ANCOVA; Difference of means in percent = 5.807, 95% CI 2-sided [-2.207 to 13.821], Standard Error of Mean 4.068; The above provided values refer to the variant "B.1.1.7 (alpha)"
Statistical Analysis 9: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.37773, ANCOVA; Difference of means in percent = 3.52, 95% CI 2-sided [-4.327 to 11.368], Standard Error of Mean 3.984; The above provided values refer to the variant "B.1.351 (beta)"
Statistical Analysis 10: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.29212, ANCOVA; Difference of means in percent = 4.413, 95% CI 2-sided [-3.821 to 12.647], Standard Error of Mean 4.18; The above provided values refer to the variant "P.1 (gamma)"
Statistical Analysis 11: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.14140, ANCOVA; Difference of means in percent = 5.961, 95% CI 2-sided [-1.998 to 13.919], Standard Error of Mean 4.04; The above provided values refer to the variant "BA.1 (omicron)"
Statistical Analysis 12: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.57090, ANCOVA; Difference of means in percent = 2.199, 95% CI 2-sided [-5.434 to 9.832], Standard Error of Mean 3.875; The above provided values refer to the variant "BA.4 (omicron)"
Statistical Analysis 13: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.11012, ANCOVA; Difference of means in percent = 6.528, 95% CI 2-sided [-1.491 to 14.548], Standard Error of Mean 4.071; The above provided values refer to the variant "BA.4.6 (omicron)"
Statistical Analysis 14: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.29755, ANCOVA; Difference of means in percent = 4.239, 95% CI 2-sided [-3.759 to 12.237], Standard Error of Mean 4.06; The above provided values refer to the variant "BA.5 (omicron)"

7. Other Pre Specified Outcome: Number of Participants With Unsolicited AEs
Description: Number of Participants with Unsolicited AEs until the end of trial
Time Frame: From Day 0 until Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B)
Number analyzed (Participants) | 25 | 27 | 135 | 135
Participants | 22 | 26 | 110 | 112

8. Other Pre Specified Outcome: Number of Participants With Solicited AEs
Description: Number of Participants with Solicited AEs for 7 days after study vaccination dose.
Time Frame: From Day 0 until Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B)
Number analyzed (Participants) | 25 | 27 | 135 | 135
Participants | 20 | 25 | 76 | 80

9. Other Pre Specified Outcome: Number of Participants With Rate of SAEs Grade ≥3
Description: Number of Participants with Rate of serious adverse events (SAEs) Grade ≥3 according to the National Cancer Institute Common Toxicity Criteria up to three months after study vaccination dose.
Time Frame: From Day 0 until Month 3
Population: Provided values refer to SAEs related to the IMP. All other trial data is available upon request.
Measure: Count of Participants; unit: Participants
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B)
Number analyzed (Participants) | 25 | 27 | 135 | 135
Participants | 0 | 0 | 1 | 0

10. Other Pre Specified Outcome: Change in Cellular Immune Response Measured by qPCR 14 Days After 4th Vaccination Dose
Description: Change in cellular immune response (CD4+ and CD8+ T cell response) to SARS-CoV-2 measured by fold change of CXCL10 mRNA levels measured by qPCR after 4th vaccination dose, to be determined in a subgroup only.
Time Frame: From Day 0 until Day 14
Population: Inclusion required completed visits at Day 0 and Day 14 with a sufficient number of aliquots as per CTP.
  Provided results are absolute values of the cellular immune response on Day 14 of tubes stimulated with peptides from spike (tube A). Samples were also stimulated with peptides from a virus membrane nucleoprotein (tube B) and with peptides from the Omicron variant (tube C). All trial results will be provided upon request.
Measure: Mean (Standard Deviation); unit: Fold change of CXCL10 mRNA levels
Groups:
- BNT162b2: vaccination with BNT162b2 as 4th vaccination
  Comirnaty(BTN162b2): Single booster shot (4th dose)
- mRNA-1273: vaccination with mRNA-1273 as 4th vaccination
  Spikevax (mRNA-1273): Single booster shot (4th dose)
Arm/Group | BNT162b2 | mRNA-1273
Number analyzed (Participants) | 79 | 92
Fold change of CXCL10 mRNA levels | 26.63 (1.58) | 26.63 (1.59)

11. Other Pre Specified Outcome: Neutralizing Antibody Titre Against Newly Emerging Variants in Bio-banked Samples After Study Vaccination Dose
Description: "Neutralizing antibody titre (Virus Neutralisation Assay)" against newly emerging variants in bio-banked samples after a 3rd (Part A) or 4th vaccination dose (Part B), to be determined in a subgroup only.
  Microneutralization assay results were proposed to be reported as "change in neutralizing antibody titre (Virus Neutralisation Assay)" in the trial protocol. However, as the pandemic progressed, the need arose to assess neutralization against different variants. In our stud(ies), we evaluated not only the Wuhan strain but also 25 distinct variants of concern (VoCs) and/or variants of interest (VoIs). For VoCs and VoIs, expressing results as "change in neutralization capacity expressed as a percentage (%)" is more effective as it illustrates the impact of mutations on neutralization, thereby allowing cross-variant comparisons. This adjustment did not alter the suggested endpoint, as both reporting methods reflect the ability of patients' antibodies neutralizing capacities.
Time Frame: From Day 0 until Month 12
Population: Titres of neutralizing antibodies were reported as change in neutralization capacity. Provided values refer to the VoI "XBB.1 (omicron)".
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B)
Number analyzed (Participants) | 21 | 20 | 120 | 120
percentage of inhibition | 19.28 (30.94) | 27.18 (28.14) | 16.75 (34.24) | 19.03 (33.01)
Statistical Analysis 1: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.39426, ANCOVA; Difference of means in percent = 9.64, 95% CI 2-sided [-12.995 to 32.275], Standard Error of Mean 11.191; The above provided values refer to the variant "P.2 (gamma)"
Statistical Analysis 2: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.42055, ANCOVA; Difference of means in percent = 8.764, 95% CI 2-sided [-13.011 to 30.539], Standard Error of Mean 10.765; The above provided values refer to the variant "B.1.617"
Statistical Analysis 3: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.44391, ANCOVA; Difference of means in percent = 8.472, 95% CI 2-sided [-13.683 to 30.627], Standard Error of Mean 10.953; The above provided values refer to the variant "B.1.617.1 (kappa)"
Statistical Analysis 4: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.43775, ANCOVA; Difference of means in percent = 8.483, 95% CI 2-sided [-13.402 to 30.368], Standard Error of Mean 10.82; The above provided values refer to the variant "AY.3 (delta)"
Statistical Analysis 5: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.53511, ANCOVA; Difference of means in percent = 6.19, 95% CI 2-sided [-13.819 to 26.2], Standard Error of Mean 9.892; The above provided values refer to the variant "AY.4.2 (delta)"
Statistical Analysis 6: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.67576, ANCOVA; Difference of means in percent = 4.552, 95% CI 2-sided [-17.295 to 26.399], Standard Error of Mean 10.801; The above provided values refer to the variant "B.1.617.3"
Statistical Analysis 7: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.45443, ANCOVA; Difference of means in percent = 8.438, 95% CI 2-sided [-14.15 to 31.027], Standard Error of Mean 11.168; The above provided values refer to the variant "B.1.526.1 (iota)"
Statistical Analysis 8: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.38904, ANCOVA; Difference of means in percent = 8.901, 95% CI 2-sided [-11.768 to 29.569], Standard Error of Mean 10.218; The above provided values refer to the variant "BA.2+L452M (omicron)"
Statistical Analysis 9: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.47466, ANCOVA; Difference of means in percent = 7.302, 95% CI 2-sided [-13.147 to 27.751], Standard Error of Mean 10.11; The above provided values refer to the variant "BA.2+L452R (omicron)"
Statistical Analysis 10: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.77110, ANCOVA; Difference of means in percent = 2.878, 95% CI 2-sided [-16.993 to 22.749], Standard Error of Mean 9.824; The above provided values refer to the variant "BA.2.12.1 (omicron)"
Statistical Analysis 11: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.86646, ANCOVA; Difference of means in percent = 1.753, 95% CI 2-sided [-19.195 to 22.701]; The above provided values refer to the variant "BA.2.75 (omicron)"
Statistical Analysis 12: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.57972, ANCOVA; Difference of means in percent = 5.42, 95% CI 2-sided [-14.21 to 25.049], Standard Error of Mean 9.705; The above provided values refer to the variant "BA.2.75.2 (omicron)"
Statistical Analysis 13: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.90166, ANCOVA; Difference of means in percent = 1.17, 95% CI 2-sided [-17.859 to 20.199], Standard Error of Mean 9.408; The above provided values refer to the variant "BA.3 (omicron)"
Statistical Analysis 14: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.92279, ANCOVA; Difference of means in percent = 1.018, 95% CI 2-sided [-20.099 to 22.136], Standard Error of Mean 10.44; The above provided values refer to the variant "BF.7 (omicron)"
Statistical Analysis 15: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.71191, ANCOVA; Difference of means in percent = 3.532, 95% CI 2-sided [-15.675 to 22.74], Standard Error of Mean 9.496; The above provided values refer to the variant "BQ.1 (omicron)"
Statistical Analysis 16: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.73415, ANCOVA; Difference of means in percent = 2.995, 95% CI 2-sided [-14.714 to 20.703], Standard Error of Mean 8.755; The above provided values refer to the variant "BQ.1.1 (omicron)"
Statistical Analysis 17: Comparison: BNT162b2 (Part A) vs mRNA-1273 (Part A); This statistical analysis reflects Part A of the study; Test type: Other; p = 0.45798, ANCOVA; Difference of means in percent = 7.157, 95% CI 2-sided [-12.155 to 26.469], Standard Error of Mean 9.548; The above provided values refer to the variant "XBB.1 (omicron)"
Statistical Analysis 18: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.23582, ANCOVA; Difference of means in percent = 4.819, 95% CI 2-sided [-3.169 to 12.808], Standard Error of Mean 4.055; The above provided values refer to the variant "P.2 (gamma)"
Statistical Analysis 19: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.19354, ANCOVA; Difference of means in percent = 5.312, 95% CI 2-sided [-2.713 to 13.337], Standard Error of Mean 4.074; The above provided values refer to the variant "B.1.617"
Statistical Analysis 20: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.17033, ANCOVA; Difference of means in percent = 5.714, 95% CI 2-sided [-2.471 to 13.899], Standard Error of Mean 4.155; The above provided values refer to the variant "B.1.617.1 (kappa)"
Statistical Analysis 21: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.13895, ANCOVA; Difference of means in percent = 5.934, 95% CI 2-sided [-1.94 to 13.808], Standard Error of Mean 3.997; The above provided values refer to the variant "AY.3 (delta)"
Statistical Analysis 22: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.26924, ANCOVA; Difference of means in percent = 4.222, 95% CI 2-sided [-3.288 to 11.732], Standard Error of Mean 3.812; The above provided values refer to the variant "AY.4.2 (delta)"
Statistical Analysis 23: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.17080, ANCOVA; Difference of means in percent = 5.49, 95% CI 2-sided [-2.382 to 13.362], Standard Error of Mean 3.996; The above provided values refer to the variant "B.1.617.3"
Statistical Analysis 24: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.18502, ANCOVA; Difference of means in percent = 5.567, 95% CI 2-sided [-2.683 to 13.818], Standard Error of Mean 4.188; The above provided values refer to the variant "B.1.526.1 (iota)"
Statistical Analysis 25: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.38344, ANCOVA; Difference of means in percent = 3.438, 95% CI 2-sided [-4.318 to 11.195], Standard Error of Mean 3.938; The above provided values refer to the variant "BA.2+L452M (omicron)"
Statistical Analysis 26: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.41100, ANCOVA; Difference of means in percent = 3.279, 95% CI 2-sided [-4.565 to 11.124], Standard Error of Mean 3.982; The above provided values refer to the variant "BA.2+L452R (omicron)"
Statistical Analysis 27: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.50660, ANCOVA; Difference of means in percent = 2.67, 95% CI 2-sided [-5.237 to 10.577], Standard Error of Mean 4.014; The above provided values refer to the variant "BA.2.12.1 (omicron)"
Statistical Analysis 28: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.28604, ANCOVA; Difference of means in percent = 4.535, 95% CI 2-sided [-3.82 to 12.891], Standard Error of Mean 4.242; The above provided values refer to the variant "BA.2.75 (omicron)"
Statistical Analysis 29: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.11715, ANCOVA; Difference of means in percent = 6.259, 95% CI 2-sided [-1.582 to 14.1], Standard Error of Mean 3.98; The above provided values refer to the variant "BA.2.75.2 (omicron)"
Statistical Analysis 30: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.33567, ANCOVA; Difference of means in percent = 3.818, 95% CI 2-sided [-3.978 to 11.613], Standard Error of Mean 3.957; The above provided values refer to the variant "BA.3 (omicron)"
Statistical Analysis 31: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.15232, ANCOVA; Difference of means in percent = 5.775, 95% CI 2-sided [-2.147 to 13.697], Standard Error of Mean 4.022; The above provided values refer to the variant "BF.7 (omicron)"
Statistical Analysis 32: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.21234, ANCOVA; Difference of means in percent = 4.808, 95% CI 2-sided [-2.766 to 12.383], Standard Error of Mean 3.845; The above provided values refer to the variant "BQ.1 (omicron)"
Statistical Analysis 33: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.22687, ANCOVA; Difference of means in percent = 4.58, 95% CI 2-sided [-2.866 to 12.026], Standard Error of Mean 3.78; The above provided values refer to the variant "BQ.1.1 (omicron)"
Statistical Analysis 34: Comparison: BNT162b2 (Part B) vs mRNA-1273 (Part B); This statistical analysis reflects Part B of the study; Test type: Other; p = 0.38832, ANCOVA; Difference of means in percent = 3.498, 95% CI 2-sided [-4.475 to 11.47], Standard Error of Mean 4.047; The above provided values refer to the variant "XBB.1 (omicron)"

ADVERSE EVENTS:
Time Frame: AEs were documented starting from baseline visit (Day 0) and until the last scheduled visit after the study vaccine dose (Month 12).
Arm/Group | BNT162b2 (Part A) | mRNA-1273 (Part A) | BNT162b2 (Part B) | mRNA-1273 (Part B)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27 | 2/135 | 5/135
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/27 | 21/135 | 22/135
Other Adverse Events (participants affected / at risk) | 20/25 | 25/27 | 103/135 | 110/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNT162b2 (Part A) (N=25) | mRNA-1273 (Part A) (N=27) | BNT162b2 (Part B) (N=135) | mRNA-1273 (Part B) (N=135)
Acute myocardial infarction (Cardiac disorders) | NA | NA | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | NA | NA | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | NA | NA | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | NA | NA | 1 (2) | 3 (4)
Atrioventricular block (Cardiac disorders) | NA | NA | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | NA | NA | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | NA | NA | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | NA | NA | 1 (2) | 1 (2)
Cardio-respiratory arrest (Cardiac disorders) | NA | NA | 1 (1) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | NA | NA | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | NA | NA | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | NA | NA | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | NA | NA | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | NA | NA | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | NA | NA | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | NA | NA | 0 (0) | 1 (1)
Chest pain (General disorders) | NA | NA | 1 (1) | 0 (0)
Chills (General disorders) | NA | NA | 1 (1) | 0 (0)
Malaise (General disorders) | NA | NA | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | NA | NA | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | NA | NA | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | NA | NA | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | NA | NA | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | NA | NA | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | NA | NA | 3 (5) | 0 (0)
Sepsis (Infections and infestations) | NA | NA | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | NA | NA | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | NA | NA | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | NA | NA | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | NA | NA | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | NA | NA | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | NA | NA | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | NA | NA | 1 (1) | 0 (0)
Femoral neck fracture (Musculoskeletal and connective tissue disorders) | NA | NA | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | NA | NA | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | NA | NA | 0 (0) | 1 (1)
Pelvic fracture (Musculoskeletal and connective tissue disorders) | NA | NA | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 (1) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 (1) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 (1) | 0 (0)
Brain stem stroke (Nervous system disorders) | NA | NA | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | NA | NA | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | NA | NA | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | NA | NA | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | NA | NA | 0 (0) | 1 (1)
Headache (Nervous system disorders) | NA | NA | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | NA | NA | 0 (0) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | NA | NA | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | NA | NA | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | NA | NA | 1 (1) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 (0) | 1 (1)
Vertebroplasty (Surgical and medical procedures) | NA | NA | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | NA | NA | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | NA | NA | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNT162b2 (Part A) (N=25) | mRNA-1273 (Part A) (N=27) | BNT162b2 (Part B) (N=135) | mRNA-1273 (Part B) (N=135)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myopic chorioretinal degeneration (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 1 (1) | 8 (9)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 14 (14) | 16 (19)
Chills (General disorders) | 1 (1) | 5 (5) | 6 (6) | 8 (8)
Discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Extensive swelling of vaccinated limb (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Fatigue (General disorders) | 7 (7) | 14 (16) | 31 (35) | 51 (57)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site dysaesthesia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 2 (3) | 4 (5) | 8 (8) | 20 (22)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 6 (6) | 10 (12) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 7 (7) | 5 (5) | 54 (55) | 59 (62)
Injection site pruritus (General disorders) | 3 (3) | 5 (5) | 9 (9) | 9 (9)
Injection site swelling (General disorders) | 2 (2) | 7 (7) | 10 (10) | 15 (15)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site vesicles (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (2) | 0 (0) | 11 (11) | 17 (18)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vaccination site movement impairment (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 31 (33) | 31 (33)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 6 (7) | 5 (5)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 3 (5)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Heart rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipids increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 4 (5) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (8) | 6 (6) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (8) | 7 (8) | 11 (11)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 34 (35) | 40 (42)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 4 (5) | 7 (7)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 5 (5) | 14 (17) | 23 (27)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Vertigo positional (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 7 (9) | 15 (17)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraphimosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 12 (14)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 12 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 3 (4) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Lens extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site discomfort (Gastrointestinal disorders) | 8 (8) | 15 (16) | 0 (0) | 0 (0)
Injection site movement impairment (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT05160766/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/66/NCT05160766/SAP_001.pdf